CLINICAL TRIAL: NCT06025435
Title: SAIA-SSP-HIV: a Systems Analysis and Improvement Approach to Optimizing HIV Service Delivery in Syringe Services Programs
Brief Title: A Systems Analysis and Improvement Approach for Optimizing HIV Service Delivery in Syringe Services Programs
Acronym: SAIA-SSP-HIV
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Drexel University (Other); RTI International (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Angela Bazzi, Associate Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 38233; R01DA056883 (NIH)
Record Dates: First submitted 2023-08-04; First posted 2023-09-06 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: HIV Infections
Keywords: Systems Analysis; Preventative Health Services; Pre-Exposure Prophylaxis; Costs and Cost Analysis; Diagnostic Screening Programs; Syringe Service Programs; Randomized Controlled Clinical Trial; Multicenter Study; Health Services Research; Facilities and Services Utilization; Retention in Care; Implementation Science; Narcotic-Related Disorders; Infectious Disease Transmission; Communicable Disease; Substance-Related Disorders
MeSH Terms: conditions — HIV Infections; Narcotic-Related Disorders; Communicable Diseases; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SAIA-SSP-HIV (Experimental): SAIA-SSP-HIV is an intervention that facilitates an organizational, SSP-level analysis of the delivery of HIV services by assigning a trained SAIA specialist to apply tools and techniques and engage staff to define barriers, identify solutions, and evaluate their success in cycles until achieving desired change regarding HIV service delivery. The scientific premise of this RCT is that SAIA will effectively boost and extend HIV service delivery cascades within SSPs assigned to the SAIA-SSP-HIV intervention condition (relative to IAU). SAIA specialists will meet with SSP staff biweekly for the first 3 months and then once monthly for the remaining 9 months during the 12-month intervention period.
  Interventions: Other: SAIA-HIV-SSP
- Implementation as usual (No Intervention): SSPs randomized to the IAU arm will not receive support from a SAIA specialist. Though many SSPs in the US already offer HIV services, the investigators are testing the ability of SAIA-SSP-HIV to optimize the delivery of HIV services within SSPs. As such, the IAU condition is characterized by the absence of SAIA-SSP-HIV with the goal of comparing whether SAIA-SSP-HIV improves SSPs' HIV service delivery cascades.

INTERVENTIONS:
Other: SAIA-HIV-SSP — The Systems Analysis and Improvement Approach (SAIA) is an evidence-based, multicomponent implementation strategy for improving the delivery of appropriate clinical services for HIV prevention and treatment. It involves five cyclical steps including (1) analyzing service delivery data to identify priority areas for system improvements, (2) mapping processes and building consensus around programmatic modifications to address priority areas, (3) implementing programmatic modifications, (4) assessing effects of programmatic modifications on improving delivery of services across the cascade, and (5) repeating steps 1-4 as needed.
  Arms: SAIA-SSP-HIV

SUMMARY:
The goal of this clinical trial is to assess the effectiveness of an evidence-based, organizational-level implementation strategy, the Systems Analysis and Improvement Approach, in improving HIV service delivery (SAIA-SSP-HIV) in U.S. syringe services programs (SSPs). The main questions it aims to answer are:

* Does SAIA-SSP-HIV improve delivery of HIV services (including the proportion of SSP participants receiving HIV testing and referrals to appropriate clinical services for HIV prevention and treatment) compared to implementation as usual (IAU)?
* Does SAIA-SSP-HIV result in sustained improvement of HIV service delivery cascades (including the proportion of SSP participants receiving HIV testing and referrals to appropriate clinical services for HIV prevention and treatment) compared to IAU?
* What are the costs associated with SAIA-SSP-HIV and how cost-effective is the strategy?

The trial will take place over 21 months and consist of a 3-month lead-in period, a 12-month active period, and a 6-month sustainment period. During the 12-month active period a SAIA specialist will meet with SSPs randomized to the SAIA-SSP-HIV arm to help them optimize their HIV service delivery cascades. Researchers will compare the SAIA-SSP-HIV and IAU arms to see if HIV service delivery and costs and cost-effectiveness differ by group.

DETAILED DESCRIPTION:
The investigators plan to examine SAIA-SSP-HIV's impact on SSPs compared to an implementation-as-usual (IAU) condition across 3 aims and several related hypotheses. Data collection will take place monthly across 21 months of SSP participation. These 21 months include a 3-month lead-in period to establish SSP outcome data characteristics, the 12-month intervention period during which sites randomized to SAIA-SSP-HIV will meet with the SAIA specialist, and an additional 6 months (sustainment period) to determine whether impacts are sustained.

* Aim 1. The first aim of the study is to assess the effectiveness of SAIA-SSP-HIV. The investigators hypothesize that compared with SSPs receiving IAU, SSPs receiving SAIA-SSP-HIV will significantly increase the proportion of SSP participants receiving HIV testing and referrals to appropriate clinical services for HIV prevention and treatment over 12 months.
* Aim 2. The second aim of the study is to assess the sustained effectiveness of SAIA-SSP-HIV. The investigators hypothesize that compared with SSPs that received IAU, SSPs that received SAIA-SSP-HIV will report a significantly higher proportion of SSP participants receiving HIV testing and referrals to appropriate clinical services for HIV prevention and treatment at 18 months.
* Aim 3. The third aim of the study is to assess the costs and cost-effectiveness of SAIA-SSP-HIV on improving HIV service delivery cascades at SSPs, relative to IAU. The investigators hypothesize that, compared to SSPs that received IAU, SSPs that received SAIA-SSP-HIV will be cost-effective at increasing the proportion of SSP participants receiving HIV testing and referrals to appropriate clinical services for HIV prevention and treatment.

To meet these aims, the investigators plan to conduct a randomized controlled interrupted time series trial among 32 U.S. SSPs (n=16 will be randomly assigned to the SAIA-SSP-HIV arm and n=16 to the IAU arm). SSPs randomized to the IAU arm will not receive support from a SAIA-SSP-HIV specialist. As such, the IAU condition is characterized by the absence of SAIA-SSP-HIV with the goal of comparing whether SAIA-SSP-HIV improves SSPs' HIV service delivery cascade.

Preliminary research has demonstrated the need for increased HIV services at SSPs and the acceptability, facilitators, and feasibility of HIV service implementation at SSPs. To the investigators' knowledge, this will be the first randomized controlled trial (RCT) of an organizational-level intervention to optimize the SSP-based HIV service delivery cascade. If successful, SAIA could be disseminated to the ≥430 SSPs nationally and in global settings, carrying the potential for exceptional impact amidst persistent HIV transmission in people who inject drugs (PWID).

The primary contact at each SSP will be asked about basic organizational characteristics (location, number of staff, budget, etc.). Next, the primary contacts as well as other staff involved with HIV service delivery at each SSP will be asked about contextual variables such as implementation climate for improving the HIV service delivery cascade. Quality control and monitoring of SAIA fidelity will include reviewing the SAIA management database for content, which will contain key information regarding SAIA specialists' delivery of the SAIA intervention to SSPs (e.g., date, service type and length, activity and name of SAIA specialist). The database will be reviewed during weekly meetings between the SAIA specialists and the study coordinator. Additionally, the SAIA specialists and study coordinator will review implementation efforts by completing periodic reflections on a monthly basis. If necessary, additional training and supervision will be conducted with the SAIA specialists. For SSPs in the SAIA arm, the investigators will routinely collect data on the number of SAIA cycles and the content and impact of programmatic changes during the active and sustainment periods to allow for observation of activities during and after SAIA delivery.

ELIGIBILITY:
Inclusion Criteria:

* Organization operates within the United States, U.S. territory, or Tribal Nation.
* Organization operates a dedicated syringe service program (SSP) that provides access to sterile syringes and injection equipment for people who inject drugs (PWID).
* In the past 30 days, SSP staff have directly provided HIV counseling and testing services to SSP participants.

Exclusion Criteria:

* Organization is participating in or has participated in other studies involving SAIA or components of SAIA.
* Organization intends to stop providing HIV counseling and testing services to SSP participants within 21 months of their respective start date.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Effectiveness | 12 months
  * 1(a) HIV Testing (Aim 1, Reach): Number of SSP participants tested for HIV, accounting for the total number of SSP participants.
  * 1(b) Total Referrals to Appropriate Clinical Services for HIV Prevention and Treatment (Aim 1, Fidelity to the cascade): Number of SSP participants referred to appropriate clinical services for HIV prevention and treatment, accounting for the number of SSP participants tested for HIV.
Sustained Effectiveness | 18 months
  * 2(a) HIV Testing (Aim 2, Reach): Number of SSP participants tested for HIV, accounting for the total number of SSP participants.
  * 2(b) Total Referrals to Appropriate Clinical Services for HIV Prevention and Treatment (Aim 2, Fidelity to the cascade): Number of SSP participants referred to appropriate clinical services for HIV prevention and treatment, accounting for the number of SSP participants tested for HIV.
Costing | 18 months
  * 3(a) Cost (Aim 3): Dollar amount of cost estimates associated with SAIA-HIV-SSP at the SSP level.
  * 3(b) Cost-Effectiveness (Aim 3): The ratio of the difference in costs to the difference in outcomes between study groups.

CONTACTS AND LOCATIONS:
Overall Officials: Alexis M Roth, PhD, Principal Investigator — Drexel University; Barrot H Lambdin, PhD, Principal Investigator — RTI International
Locations (1):
- University of California, San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maki M, Jarvinen N, Rabina J, Roos C, Maaheimo H, Renkonen R; Pirkko; Mattila. Functional expression of Pseudomonas aeruginosa GDP-4-keto-6-deoxy-D-mannose reductase which synthesizes GDP-rhamnose. Eur J Biochem. 2002 Jan;269(2):593-601. doi: 10.1046/j.0014-2956.2001.02688.x. PMID 11856318
- [Background] Bazzi AR, Biancarelli DL, Childs E, Drainoni ML, Edeza A, Salhaney P, Mimiaga MJ, Biello KB. Limited Knowledge and Mixed Interest in Pre-Exposure Prophylaxis for HIV Prevention Among People Who Inject Drugs. AIDS Patient Care STDS. 2018 Dec;32(12):529-537. doi: 10.1089/apc.2018.0126. Epub 2018 Oct 11. PMID 30311777
- [Background] Biello KB, Bazzi AR, Vahey S, Harris M, Shaw L, Brody J. Delivering Preexposure Prophylaxis to People Who Use Drugs and Experience Homelessness, Boston, MA, 2018-2020. Am J Public Health. 2021 Jun;111(6):1045-1048. doi: 10.2105/AJPH.2021.306208. PMID 33950728
- [Background] Biello KB, Bazzi AR, Mimiaga MJ, Biancarelli DL, Edeza A, Salhaney P, Childs E, Drainoni ML. Perspectives on HIV pre-exposure prophylaxis (PrEP) utilization and related intervention needs among people who inject drugs. Harm Reduct J. 2018 Nov 12;15(1):55. doi: 10.1186/s12954-018-0263-5. PMID 30419926
- [Background] Biello KB, Mimiaga MJ, Valente PK, Saxena N, Bazzi AR. The Past, Present, and Future of PrEP implementation Among People Who Use Drugs. Curr HIV/AIDS Rep. 2021 Aug;18(4):328-338. doi: 10.1007/s11904-021-00556-z. Epub 2021 Apr 27. PMID 33907971
- [Background] Brody JK, Taylor J, Biello K, Bazzi AR. Towards equity for people who inject drugs in HIV prevention drug trials. Int J Drug Policy. 2021 Oct;96:103284. doi: 10.1016/j.drugpo.2021.103284. Epub 2021 Jun 3. No abstract available. PMID 34092469
- [Background] Earlywine JJ, Bazzi AR, Biello KB, Klevens RM. High Prevalence of Indications for Pre-exposure Prophylaxis Among People Who Inject Drugs in Boston, Massachusetts. Am J Prev Med. 2021 Mar;60(3):369-378. doi: 10.1016/j.amepre.2020.09.011. Epub 2020 Nov 21. PMID 33229144
- [Background] Edeza A, Bazzi A, Salhaney P, Biancarelli D, Childs E, Mimiaga MJ, Drainoni ML, Biello K. HIV Pre-exposure Prophylaxis for People Who Inject Drugs: The Context of Co-occurring Injection- and Sexual-Related HIV Risk in the U.S. Northeast. Subst Use Misuse. 2020;55(4):525-533. doi: 10.1080/10826084.2019.1673419. Epub 2019 Oct 9. PMID 31596171
- [Background] Felsher M, Ziegler E, Smith LR, Sherman SG, Amico KR, Fox R, Madden K, Roth AM. An Exploration of Pre-exposure Prophylaxis (PrEP) Initiation Among Women Who Inject Drugs. Arch Sex Behav. 2020 Aug;49(6):2205-2212. doi: 10.1007/s10508-020-01684-0. Epub 2020 Apr 9. PMID 32274742
- [Background] Roth AM, Tran NK, Felsher M, Gadegbeku AB, Piecara B, Fox R, Krakower DS, Bellamy SL, Amico KR, Benitez JA, Van Der Pol B. Integrating HIV Preexposure Prophylaxis With Community-Based Syringe Services for Women Who Inject Drugs: Results From the Project SHE Demonstration Study. J Acquir Immune Defic Syndr. 2021 Mar 1;86(3):e61-e70. doi: 10.1097/QAI.0000000000002558. PMID 33148998
- [Derived] Bazzi AR, Roth AM, Akiba CF, Huffaker SL, Patel SV, Smith J, Laurano R, Orme S, Zarkin GA, Morgan-Lopez A, Lambdin BH. A systems analysis and improvement approach to optimizing syringe services programs' delivery of HIV testing and referrals: Study protocol for a parallel-group randomized controlled trial (SAIA-SSP-HIV). PLoS One. 2025 Feb 25;20(2):e0319340. doi: 10.1371/journal.pone.0319340. eCollection 2025. PMID 39999129